CLINICAL TRIAL: NCT00988416
Title: PET-CT for Intraductal Papillary Mucinous Neoplasm (IPMN)
Brief Title: Positron Emission Tomography-computed Tomography (PET-CT) for Main & Branch Intraductal Papillary Mucinous Neoplasm
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Christian M. Schmidt, Professor of Surgery, Biochemistry and Molecular Biology, Indiana University
Other Study IDs: 0810-11
Record Dates: First submitted 2009-09-29; First posted 2009-10-02 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Intraductal Papillary Mucinous Neoplasm
Keywords: IPMN

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: PET-CT — Pancreas Protocol PET-CT

SUMMARY:
The purpose of the study is to prove the hypothesis that pancreas PET-CT can differentiate duct involved IPMN with malignancy from duct involved non-malignant IPMN.

DETAILED DESCRIPTION:
Duct involved intraductal papillary mucinous neoplasm is associated with a 35-70% (particularly involving the main duct) incidence of malignancy. Current guidelines recommend pancreatic resection for fit patients with main or branch duct involved IPMN. Pancreatic resection can be associated with morbidity and mortality. Reliable tests or biomarkers accurately differentiating non-malignant from malignant duct involved IPMN are non-existent. Test or biomarkers differentiating duct involved from duct uninvolved IPMN are also inaccurate. Patients with suspected duct IPMN with symptoms have a higher chance of associated malignancy. These findings are not specific for malignant IPMN so, if relied on, they would results in missed malignancies as well as potentially unnecessary operations in a significant percentage of patients. PET scanning has been studied retrospectively and purported to be a highly reliable indicator og high grade dysplasia and/or invasive cancer in patients with IPMN. Thus, PET could represent a future standard of care by some authorities in the work-up of patients with IPMN. This proposal seeks to prove the hypothesis that pancreas PET-CT can differentiate duct involved IPMN with malignancy from duct involved IPMN without malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for the study if they have a clinical and/or cytopathologic diagnosis of IPMN (primary or recurrent) with suspected main or branch duct involvement.
* A clinical diagnosis of IPMN with main duct involvement will be determined by the surgeon caring for the patient. Main duct involvement may be suspected where there is a significant radiographic character change (cystic dilation) in the main pancreatic duct (independent of ductal diameter), a significant "step-up" in main duct diameter (2-3 fold) or a significant segmental or diffuse dilation of the main pancreatic duct (> or equal to 4mm) as defined by CT, MRCP, EUS or ERCP.
* All patients with a diagnosis (pathologic) or presumed diagnosis (based upon clinical presentation) of IPMN and who are to undergo surgical treatment are eligible for the study. This may include patients who have already undergone IPMN surgery in the past and who are expected to undergo a second IPMN surgery.
* Patients with unrecoverable renal function on dialysis are eligible to undergo this study.
* Female patients of child-bearing age must have a negative urine or serum pregnancy test prior to enrollment.
* Subjects must have medical insurance or Medicare willing to pay for the cost of this PET-CT procedure or the CT portion of the procedure.

Exclusion Criteria:

* Patients who despite suspected duct involved IPMN are not fit surgical candidates and thus will not undergo resection of their IPMN.
* Patients with uncontrolled serum glucose will not be eligible for the study due to the unreliability of PET in these patients. Diabetic patients are eligible as long as their glucose is reasonably controlled (as determined by the nuclear medicine radiologists). The Department of Radiology has a Standard Operating Procedure in place for the management of these patients which will be followed in this protocol.
* Pediatric patients are excluded from this study since IPMN is a diagnosis present in adult patients.
* Female patients who are pregnant or who are currently breastfeeding.
* Patients with allergy to IV contrast have a relative contraindication to the study. Some of these patients at the discretion of the investigator may undergo a standard protocol of pre-IV contrast steroids to manage their allergic response. The Department of Radiology has guidelines that will be followed in this protocol for patients who have experienced an allergic reaction to IV contrast.
* Patients with renal insufficiency (creatinine > or equal to 2.0) have a relative contraindication to the study. At the investigator's discretion these patients may be enrolled and undergo PET-CT without IV contrast.
* Patients without insurance or Medicare coverage or patients with insurance/Medicare coverage but insurer is unwilling to pay for the cost of the PET-CT procedure or the CT portion of the procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are selected from group of patients in whom IPMN is suspected as they are seen in the clinic for consultation with the surgeon regarding their surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2009-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pancreas PET-CT can differentiate duct involved IPMN with malignancy from duct involved IPMN without malignancy. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Christian M Schmidt, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Medical Center, Indianapolis, Indiana, United States